CLINICAL TRIAL: NCT05127772
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Ascending Single and Multiple Doses to Evaluate the Safety, Tolerability, PK, PDand Randomized, Open-label，Crossover, Food Effect Study of HEC93077 in Healthy Chinese Subjects and Hyperuricemia Patients
Brief Title: A Clinical Trial of HEC93077 in Chinese Healthy Subjects and HUA Patients With Single or Multiple Dosing
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC93077-HUA-101
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- single dose of HEC93077（pilot trial arm） (Experimental): Healthy subjects receive single dose of HEC93077
  Interventions: Drug: HEC93077
- single dose of HEC93077（Cohort 1） (Experimental): Healthy subjects receive sinele dose of HEC93077 or matching placebo
  Interventions: Drug: HEC93077; Drug: Placebo
- single dose of HEC93077（Cohort 2） (Experimental): Healthy subjects receive sinele dose of HEC93077 or matching placebo
  Interventions: Drug: HEC93077; Drug: Placebo
- single dose of HEC93077（Cohort 3,Fed/Fasting） (Experimental): Following an overnight fast of at least 10 hours, a single dose of HEC93077 or placebo will be administered on 2 separate occasions (fasting and after meal) in a randomized crossover fashion with different food restrictions.
  Interventions: Drug: HEC93077; Drug: Placebo
- single dose of HEC93077（Cohort 4） (Experimental): Healthy subjects receive sinele dose of HEC93077 or matching placebo
  Interventions: Drug: HEC93077; Drug: Placebo
- single dose of HEC93077（Cohort 5） (Experimental): Healthy subjects receive sinele dose of HEC93077 or matching placebo
  Interventions: Drug: HEC93077; Drug: Placebo
- single dose of HEC93077（Cohort 6） (Experimental): Healthy subjects receive sinele dose of HEC93077 or matching placebo
  Interventions: Drug: HEC93077; Drug: Placebo
- single dose of HEC93077（Cohort 7） (Experimental): Healthy subjects receive sinele dose of HEC93077 or matching placebo
  Interventions: Drug: HEC93077; Drug: Placebo
- multiple doses of HEC93077（ Cohort 8） (Experimental): Healthy subjects receive multiple doses of HEC93077 or matching placebo
  Interventions: Drug: HEC93077; Drug: Placebo
- multiple doses of HEC93077（ Cohort 9, Group 1) (Experimental): Healthy subjects receive multiple doses of HEC93077 or matching placebo
  Interventions: Drug: HEC93077; Drug: Placebo
- multiple doses of HEC93077（ Cohort 9, Gruop 2) (Experimental): Hyperuricemia subjects receive multiple doses of HEC93077 or matching placebo
  Interventions: Drug: HEC93077; Drug: Placebo
- multiple doses of HEC93077（ Cohort 10) (Experimental): Healthy subjects receive multiple doses of HEC93077 or matching placebo
  Interventions: Drug: HEC93077; Drug: Placebo

INTERVENTIONS:
Drug: HEC93077 — Paticipants recieve HEC93077 orally single or Mulltiple doses up to 14 days
Drug: Placebo — Paticipants recieve placebo matching HEC93077 orally single or Mulltiple doses up to 14 days
  Arms: multiple doses of HEC93077（ Cohort 10); multiple doses of HEC93077（ Cohort 8）; multiple doses of HEC93077（ Cohort 9, Group 1); multiple doses of HEC93077（ Cohort 9, Gruop 2); single dose of HEC93077（Cohort 1）; single dose of HEC93077（Cohort 2）; single dose of HEC93077（Cohort 3,Fed/Fasting）; single dose of HEC93077（Cohort 4）; single dose of HEC93077（Cohort 5）; single dose of HEC93077（Cohort 6）; single dose of HEC93077（Cohort 7）

SUMMARY:
A phase 1 clinical trial of HEC93077,to evaluate the safety ,PK,PD and food effect in Chinese healthy subjects and HUA patients after single or multiple dosing.

ELIGIBILITY:
Healthy Subjects：

Inclusion Criteria:

1. Subjects who are willing and are able to provide a written informed consent to participate in the study.
2. Subjects aged between 18 and 45 (both inclusive) years old.
3. Healthy volunteers has a body weight ≥50 kg (for male) or ≥ 45kg (for female) and body mass index ≥19 and ≤28 kg/m2 at screening.
4. Subjects, who are healthy, as having no clinically significant abnormalities in vital signs, physical examination, clinical laboratory test results, Chest X-ray and 12-lead electrocardiogram (ECG).
5. Without Plan for pregnancy or pregnant within 3 months after enrollment throughout the trial.
6. Serum uric acid≥240 and<420 at screening.
7. GFR≥90 mL/min/1.73 m2 at screening.

Exclusion Criteria:

1. At screening subjects have the following diseases of clinical significance, including but not limited to cardiovascular system diseases, digestive system diseases, respiratory system diseases, urinary system diseases, endocrine and metabolic system diseases, blood system diseases, central nervous system and/or mental system diseases, immune system diseases, tumors, etc.
2. A history of gastrointestinal, liver, or kidney disease or surgery prior to screening that could potentially affect the absorption, distribution, metabolism, and excretion of the test drug (except for uncomplicated appendectomy and hernia repair);
3. History of urolithiasis or ultrasound screening showed urolithiasis, renal/ureteral malformation, unirenal or renal atrophy, polycystic kidney and other urological diseases
4. History of gout and/or hyperuricemia
5. Acute illness or concomitant use from signing the ICF to initial dosing.
6. Known allergic reactions or hypersensitivity to any excipient of the drug formulation(s)， anaphylaxis physique.(Allergic to more than 3 foods and/or medications)
7. History of alcoholism or drink regularly within 3 months prior to the study(defined as Alcohol consumption of > 21 units/week), or positive results from alcohol breath test at screening.
8. History of drug abuse, or use of drugs within 2 years prior to the study,or positive results from urine drug screen test at screening.
9. Regular smoking of more than 10 cigarettes per day within 3 months before screening period, or inability to refrain from smoking during the course of the study after signing ICF.
10. Subjects with a positive serology for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies and/or TP antibodies at screening.
11. Use of any prescription or non-prescription medications、vitamin and traditional Chinese medicine within 2 weeks prior to initial dosing,or use of any mediciations which affect UA synthesize,metabolize and excrete within 4 weeks prior to initial dosing.
12. Use of any medications known to strongly inhibit and/or induce cytochrome P enzyme drug metabolism within 4 weeks prior to initial dosing.
13. Have taken any food or drink that affects CYP3A4 and/or CYP1A2 metabolic enzymes within 2 days prior to initial dosing,such as grapefruit or grapefruit drink.
14. Have taken chocolate, any food or drink containing caffeine or rich in xanthine within 72 hours prior to initial dosing.
15. Have taken any alcoholic product within 48 hours prior to initial dosing.
16. Donate blood or lose blood 400 mL or more within 1 month prior to initial dosing.
17. Subjects who plan to receive or have had organ transplants.
18. Females who are lactating/breastfeeding, or positive result from pregnancy test for women of child-bearing potential.
19. Subjects who participated in another clinical trial within 3 months prior to initial dosing.
20. Subjects who canot tolerate fat food.(only suitable to FE trial)
21. Subjects who maynot complete for other reasons.
22. Any other condition with in the opinion of the investigator would render the patient unsuitable for inclusion in the study.

Hyperuricemia Patients：

Inclusion Criteria:

1. Patients who are willing and are able to provide a written informed consent to participate in the study.
2. Patients aged between 18 and 60 (both inclusive) years old.
3. Patients has a body weight ≥50 kg (for male) or ≥ 45kg (for female) and body mass index ≥19 and ≤30 kg/m2 at screening.
4. During screening period, serum uric acid was ≥480 µmol/L twice on different days.Patients are considered to need to lower UA with a long term therapy;
5. Without Plann for pregnancy or pregnant within 3 months after enrollment throughout the trial.
6. GFR≥90 mL/min/1.73 m2 at screening.

Exclusion Criteria:（mainly different with healthy subjects）

1. Patients with myocardial infarction, angina pectoris, percutaneous coronary angioplasty, coronary artery bypass grafting, cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage or transient ischemic attack within 6 months prior to screening.
2. History of acute gout attack prior to initial dosing;
3. Acute illness or use of a contraindicated drug under the protocol from signing the ICF to initial dosing.
4. At screening,AST or ALT or TBIL >1.2 × ULN, or sCr >ULN，or HbA1c>8%.

4.Investigator judged the following conditons unsuitable for inclusion:Medical history, physical examination, electrocardiogram, chest X-ray, ultrasonic examination of digestive system , ultrasonic examination of urinary system and laboratory examination have abnormal and clinical significance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2023-10-25 (Estimated); Study Completion 2023-11-25 (Estimated)

PRIMARY OUTCOMES:
the Number of Adverse Events (AEs) | up to 25 days
  To investigate the safety and tolerability by assement of AEs following administration of oral solution in SAD and MAD
PK parameters - AUC0-∞ | up to 18 days
  Area Under the Curve(AUC)
PK parameters - Cmax | up to 18 days
  Geometric Mean of Maximum Observed Plasma Concentration of HEC93077
PK parameters -tmax | up to 18 days
  maximum observed plasma concentration
PK parameters -t½ | up to 18 days
  apparent terminal elimination half-life
PK parameters -Vz/F | up to 18 days
  apparent volume of distribution
PD parameters | up to 18 days
  Percentage of serum uric acid changed from baseline
PK parameters - Ae0-t(urine) | up to 18 days
  The amount of drug excreted in the urine
PK parameters - Ae0-t(feces) | up to 18 days
  The amount of drug excreted in the feces
PK parameters-The cumulative rate of excretion | up to 18 days
  The cumulative rate of durg excreted through urine/feces

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Universicity Care of Luzhong Hospital, Zibo, Shandong, China

IPD SHARING:
Plan to Share IPD: No